CLINICAL TRIAL: NCT02081937
Title: Anti-CD19 Chimeric Antigen Receptor Modified T Cells Infusion in Mantle Cell Lymphoma
Brief Title: CART-19 Immunotherapy in Mantle Cell Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Quanshun Wang, Dr., Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN301-XYK-CAR001
Record Dates: First submitted 2014-03-06; First posted 2014-03-07 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Hematopoietic/Lymphoid Cancer; Non-hodgkin Lymphoma,B Cell; Mantle Cell Lymphoma
Keywords: chimeric antigen receptor; immunotherapy; T lymphocyte; mantle cell lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anti-CD19 CAR T cells (Experimental): Patients receive anti-CD19-CAR retroviral vector-transduced autologous or donor-derived T cells on d1-5 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: anti-CD19-CAR vector-transduced T cells

INTERVENTIONS:
Biological: anti-CD19-CAR vector-transduced T cells
  Other Names: Genetically engineered lymphocyte therapy

SUMMARY:
Patients receive anti-CD19-CAR (coupled with CD137 and CD3 zeta signalling domains)vector-transduced autologous T cells over a period of 4 or 5 consecutive days in an escalating dose. After completion of study treatment, patients are followed intensively for 6 months, every 3 months for 2 years, and annually thereafter for 10 years.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and efficacy of the chimeric antigen receptor T cells transduced with the anti-CD19 (cluster of differentiation antigen 19 ) vector (referred to as CART-19 cells) in elderly patients with MCL.

II. Determine duration of in vivo survival of CART-19 cells. RT-PCR (reverse transcription polymerase chain reaction) analysis of whole blood will be used to detect and quantify survival of CART-19 TCR (T-cell receptor) zeta:CD137 and TCR zeta cells over time.

SECONDARY OBJECTIVES:

For patients with detectable disease, measure anti-tumor response due to CART-19 cell infusions.

Estimate relative trafficking of CART-19 cells to tumor in bone marrow and lymph nodes.

Determine if cellular or humoral host immunity develops against the murine anti-CD19, and assess correlation with loss of detectable CART-19 (loss of engraftment).

ELIGIBILITY:
Inclusion Criteria:

* Male and female with CD19+ relapsed or refractory MCL, and with no available curative treatment options (such as autologous or allogeneic SCT) who have limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled.
* Not eligible or appropriate for conventional allogeneic SCT
* Patients who achieve only a partial response to FCR(fludarabine, cyclophosphamide and Rituxan) as initial therapy will be eligible.
* Beyond 1st CR (complete remission) with relapsed or persistent disease and not eligible or appropriate for conventional allogeneic or autologous SCT
* Disease responding or stable after most recent therapy (chemotherapy, MoAb, etc...)
* Relapsed after prior autologous SCT
* Residual disease after primary therapy and not eligible for autologous SCT
* Relapsed after prior autologous SCT
* Beyond 1st CR with relapsed or persistent disease and not eligible or appropriate of conventional allogeneic or autologous SCT
* Expected survival > 12 weeks
* Creatinine < 2.5 mg/dl
* ALT(alanine aminotransferase)/AST (aspartate aminotransferase)< 3x normal
* Bilirubin < 2.0 mg/dl
* Any relapse after prior autologous SCT will make patient eligible regardless of other prior therapy
* Adequate venous access for apheresis, and no other contraindications for leukapheresis
* Voluntary informed consent is given

Exclusion Criteria:

* • Pregnant or lactating women. The safety of this therapy on unborn children is not known. Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion.
* Uncontrolled active infection
* Active hepatitis B or hepatitis C infection
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
* Previously treatment with any gene therapy products
* Feasibility assessment during screening demonstrates < 30% transduction of target lymphocytes, or insufficient expansion (< 5-fold) in response to CD3/CD137 costimulation
* Any uncontrolled active medical disorder that would preclude participation as outlined
* HIV infection

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | Until 2 years
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to the study.

SECONDARY OUTCOMES:
Clinical responses to CART-19 cell therapy | Until 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology of Chinese PLA General Hospital, Beijing, Beijing Municipality, China